CLINICAL TRIAL: NCT00627029
Title: Evaluation of Programs of Coordinated Care and Disease Management
Acronym: Coca
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MPR 8756; CMS 500-95-0047(09
Record Dates: First submitted 2008-02-15; First posted 2008-02-29 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Congestive Heart Failure; Diabetes; Coronary Artery Disease; Chronic Obstructive Pulmonary Disease; Cancer; Cerebrovascular Disease; Alzheimer's Disease; Psychotic Disorder; Major Depression
Keywords: Care coordination; Disease management; Medicare; Fee-for-service; Random assignment; Elderly
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive; Neoplasms; Cerebrovascular Disorders; Alzheimer Disease; Psychotic Disorders; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Care coordination, consisting variously (depending on the demonstration site)--nurse telephonic counseling, nurse in-person home visits, home telemonitoring equipment, and physician education and feedback.
  Interventions: Behavioral: Care Coordination
- Control (No Intervention): Usual care in Medicare fee-for-service from beneficiaries' physicians and other health care providers

INTERVENTIONS:
Behavioral: Care Coordination — Depending on the demonstration site, may consist of nurse telephonic counseling and monitoring, nurse in-person or home visits, home telemonitoring equipment, patient educational materials, patient group educations classes, physician education and feedback.
  Arms: Intervention

SUMMARY:
This is a Congressionally mandated study. In the original study, 16 demonstration programs provided care coordination services to beneficiaries with chronic illness in Medicare's fee-for-service program. A five-year CMS-funded study tested whether the programs can improve patients' use of medical services, improve patients' outcomes and satisfaction with care, and reduce Medicare costs. The study also assessed physicians' satisfaction with the programs.

In 2008 Congress extended the project for two of the original programs--Mercy Medical Center - North Iowa and Health Quality Partners in Pennsylvania--and they will enroll Medicare beneficiaries and provide care coordination services into the spring of 2010.

DETAILED DESCRIPTION:
Mathematica Policy Research, Inc. (MPR) evaluated 16 independent demonstration sites that provide coordinated care interventions to Medicare beneficiaries with chronic illnesses. The rationale for the demonstration is the lack of coordination among the multiple providers typically serving Medicare beneficiaries with chronic illnesses, as well as the adverse consequences of the lack of coordination for the beneficiaries and for Medicare costs. The demonstration sites, selected in early 2001, offered programs designed to improve both the care that patients receive and patients' knowledge of, and adherence with, recommended self-care and behavior. The study estimated the effects of each site on patients' well-being and satisfaction, in addition to the site's effects on the use and cost of Medicare covered services. This analysis relied on a patient survey conducted 6 to 12 months after enrollment, and on Medicare claims data and any data available from the demonstration sites that could enhance the study. The study included two rounds of physician surveys. In each site, eligible applicants were randomly assigned to treatment and control groups. An extensive process analysis was conducted to describe the interventions in detail, with the key goal being an assessment of those factors that account for program success and failure. The study included case studies of each site, program profiles, interim site-specific memos, two interim summary reports, two reports to Congress (based on the interim summary reports), and a final summary report. This original study enrolled 18,277 beneficiaries.

In 2008 Congress extended the study for 2 of the sites, Mercy Medical Center - North Iowa and Health Quality Partners in Pennsylvania, and they will recruit beneficiaries and provide demonstration intervention services through the spring of 2010. Mathematica Policy Research will evaluate the results of this extended demonstration using Medicare claims data and qualitative site visits to the two programs.

ELIGIBILITY:
Inclusion Criteria:

* Meets clinical and prior health service use criteria of each of the 16 demonstration sites (vary across demonstration programs)
* Resides in catchment area of one of the programs
* Enrolled in Medicare fee-for-service program
* Coverage by both Medicare Parts A and B
* Medicare is primary payer

Exclusion Criteria:

* Does not meet any of the relevant program's exclusion criteria (vary across demonstration programs)
* Not enrolled in a Medicare Advantage plan (Medicare managed care program)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18277 (Actual)
Dates: Start 2000-09; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Medicare program expenditures | Eight years

SECONDARY OUTCOMES:
Claims-based and patient-reported quality of care | Eight years

CONTACTS AND LOCATIONS:
Overall Officials: Randall S. Brown, Ph.D., Study Director — Mathematica Policy Research, Inc.; Carol A. Magee, Ph.D., Study Director — Centers for Medicare & Medicaid Services
Locations (15):
- United States (15):
  - Hospice of the Valley MediCaring Project, Phoenix, Arizona
  - Georgetown University Medical Center-Mind My Heart Program, Washington D.C., District of Columbia
  - Quality Oncology/Matria Healthcare, Sunrise, Florida
  - CorSolutions/Matria Healthcare, Rosemont, Illinois
  - Carle Foundation and Hospital, Urbana, Illinois
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Medical Care Development, Augusta, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Charlestown/Erickson Retirement Communities, Catonsville, Maryland
  - Washington University-St.Louis School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri
  - QMed, Inc., Eatontown, New Jersey
  - Lovelace Health Systems, Albuquerque, New Mexico
  - Jewish Home Lifecare, New York, New York
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - CenVaNet, Richmond, Virginia

REFERENCES:
- [Derived] Peikes D, Chen A, Schore J, Brown R. Effects of care coordination on hospitalization, quality of care, and health care expenditures among Medicare beneficiaries: 15 randomized trials. JAMA. 2009 Feb 11;301(6):603-18. doi: 10.1001/jama.2009.126. PMID 19211468
- See also: The Evaluation of the Medicare Coordinated Care Demonstration: Findings for the First Two Years — http://www.cms.hhs.gov/reports/downloads/Brown.pdf